CLINICAL TRIAL: NCT01600040
Title: Pilot Study of Adjuvant Proton Beam Teletherapy for Post-Hysterectomy Cancers of the Uterus and Cervix With Metastases to Regional Lymph Nodes
Brief Title: Proton Beam Teletherapy for Post-Hysterectomy Cancers of the Uterus and Cervix
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Andrea Russo, MD, Director, Gynecologic Radiation Oncology, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10-269
Record Dates: First submitted 2012-05-14; First posted 2012-05-16 (Estimated); Results first posted 2024-10-29 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Uterine Cancer; Cervical Cancer
Keywords: metastatic
MeSH Terms: conditions — Uterine Neoplasms; Uterine Cervical Neoplasms; Neoplasm Metastasis | interventions — Protons

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Proton Radiation Therapy (Other): This is a single arm study; all participants will receive proton radiation therapy.
  Interventions: Radiation: Proton radiation therapy

INTERVENTIONS:
Radiation: Proton radiation therapy — 5 days per week (Mon-Fri) for 5-6 weeks

SUMMARY:
Proton beam radiation therapy is known to spare surrounding normal tissues from radiation. Proton beam radiation delivers less radiation beyond the area of the target tissues. This may reduce side effects that patients would normally experience with standard (photon) radiation therapy which tends to unavoidably include more normal tissue along with tumor target tissue.

In this research study, the investigators are looking to determine if proton beam radiation is effective in controlling your cancer growth. The investigators are also looking to see if proton beam radiation can reduce side effects when compared to standard radiation treatment (photon radiation).

DETAILED DESCRIPTION:
Subjects will receive proton beam radiation treatment as an outpatient at the Francis H. Burr Proton Center at Massachusetts General Hospital, 5 days per week (Mon-Fri) over 5-6 weeks depending on the type of cancer.

Tests and procedures during study treatment (weekly):

* Questions about health and current medications
* Physical exam, includes height, weight and vital signs
* Performance status
* Blood test for complete blood counts and blood clotting (2 tsps). Repeated twice weekly for uterine cancer subjects and once weekly for cervix cancer subjects
* Pelvic exam (at week 6 only)
* Quality of life questionnaires

After completion of proton beam radiation treatment, subjects will be followed for 5 years. Follow-up visits will occur every 3 months for 2 years; every 4 months to year 3 and every 6 months thereafter. At each visit subjects will receive:

* A medical history
* Physical exam
* Performance status
* Pelvic exam
* CT scan of the chest, abdomen and pelvis every 6 months to year 3
* Quality of life questionnaires (6, 12, 24, 36, 48, and 60 months)

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed primary cancer of the uterus or cervix with histologically confirmed metastasis to one or more parametrial, pelvic or paraaortic nodes prior to enrollment. Subjects diagnosed at other institutions must have pathology reviewed and confirmed at MGH or another DF/HCC institution
* Have undergone simple, modified radical, or radical abdominal hysterectomy or vaginal hysterectomy and lymphadenectomy by open or laparoscopic assisted technique
* Life expectancy greater than 18 months
* Adequate organ and bone marrow function
* Uterine cancer subjects will be FIGO stage IIIC and may have endometrioid cancer, clear cell cancer, uterine papillary serous cancer, carcinosarcoma, or endometrial stromal sarcoma
* Cervical cancer subjects will be AJCC stages pT1,2,N1,M0 with squamous carcinoma, adenocarcinoma, adenosquamous carcinoma, or glassy cell carcinoma histology
* ECOG performance status ≤ 2 or Karnofsky performance status ≥ 60%

Exclusion Criteria:

* Prior therapeutic radiation exposure to target tissues for protocol radiation
* Evidence of extra-abdominal cancer dissemination or hematogenous cancer dissemination
* Evidence of measurable residual disease following hysterectomy and lymphadenectomy
* History of a different malignancy except if disease-free for at least 5 years and are deemed by the investigator ro be at low risk for recurrence of that malignancy. Subjects with the following cancers are eligible if diagnosed and treated within the past 5 years: cervical cancer in situ, and basal cell or squamous cell carcinoma of the skin

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2013-08 (Actual); Primary Completion 2022-10-19 (Actual); Study Completion 2023-08-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Russo, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Proton Radiation Therapy
Started | 22
Completed | 21
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: 22 patients enrolled, and 1 patient withdrew consent prior to study treatment. The other 21 patients were included in the final analyses.
Arm/Group | Proton Radiation Therapy
Number analyzed (Participants) | 21
Age, Continuous [Median (Full Range); unit: years] | 59.7 [31.5 to 79.2]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 19
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 21
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Dosimetric Comparison of Proton Beam Treatment With 3-dimensional Conformal Radiation Therapy (3DCRT) and Intensity Modulated Radiation Therapy (IMRT)
Description: In a population of women with cancers of the cervix or endometrium with pathologically proven spread to regional lymph nodes, dose volume histograms (DVH) were compared between scanning proton beam teletherapy, 3-dimensional conformal radiation therapy (3DCRT) and intensity modulated radiation therapy (IMRT). Structure sets contoured for the proton beam therapy delivered on study were used to plan alternative 3DCRT and IMRT plans by the the same medical physics team (3DCRT and IMRT were not used on study; actual dose for proton beam was compared to the doses that would have been delivered for 3DCRT or IMRT.)
  Median, 25th percentile, and 75th percentile doses are listed below by tissue volume irradiated (mL) or percentage irradiated (%) for each modality. Dose is measured in grays (Gy), which is defined as the absorption of one joule of radiation energy per kilogram of matter.
Time Frame: 5 years
Population: 22 patients enrolled, 1 of whom withdrew consent prior to study treatment. Remaining 21 patients were included in the final analysis.
Measure: Median (Inter-Quartile Range); unit: Gy
Arm/Group | Proton Radiation Therapy
Number analyzed (Participants) | 21
Gy
  3DCRT: Bowel V45 (mL) | 455.0 [361.0 to 597.0]
  IMRT: Bowel V45 (mL) | 149.0 [112.0 to 269.0]
  Proton Beam: Bowel V45 (mL) | 202.0 [132.0 to 270.0]
  3DCRT: Bowel V40 (mL) | 639.0 [492.0 to 757.0]
  IMRT: Bowel V40 (mL) | 464.0 [291.0 to 552.0]
  Proton Beam: Bowel V40 (mL) | 395.0 [299.0 to 444.0]
  3DCRT: Bowel V30 (mL) | 819.0 [663.0 to 1316.0]
  IMRT: Bowel V30 (mL) | 818.0 [640.0 to 1085.0]
  Proton beam: Bowel V30 (mL) | 536.0 [488.0 to 644.0]
  3DCRT: Bowel V20 (mL) | 2076.0 [1404.0 to 2284.0]
  IMRT: Bowel V20 (mL) | 1480.0 [1053.0 to 1915.0]
  Proton beam: Bowel V20 (mL) | 696.0 [622.0 to 833.0]
  3DCRT: Bone marrow V20 (%) | 78.4 [72.1 to 82.2]
  IMRT: Bone marrow V20 (%) | 64.0 [58.8 to 70.2]
  Proton beam: Bone marrow V20 (%) | 60.7 [55.8 to 65.1]
  3DCRT: Bone marrow V10 (%) | 85.3 [80.4 to 89.3]
  IMRT: Bone marrow V10 (%) | 64.0 [58.8 to 70.2]
  Proton beam: Bone marrow V10 (%) | 60.7 [55.8 to 65.1]
  3DCRT: Kidney V14 (%) | 30.8 [7.4 to 47.4]
  IMRT: Kidney V14 (%) | 22.1 [6.9 to 28.2]
  Proton beam: Kidney V14 (%) | 18.2 [2.7 to 25.2]

2. Primary Outcome: Acute Radiation Side Effects
Description: Acute radiation side effects were prospectively assessed. Below are the treatment-related acute toxicities (adverse events possibly, probably, or definitely related to protocol treatment that started within 4 weeks of treatment completion) that occurred on study, along with the number of participants who experienced each event at a given severity (Grade 1/mild, Grade 2/moderate, Grade 3/severe) according to the CTCAE v 4.02 (Common terminology criteria for adverse events).
Time Frame: 10 weeks
Population: 22 patients enrolled, 1 of whom discontinued prior to study treatment. The remaining 21 patients were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Proton Radiation Therapy
Number analyzed (Participants) | 21
Participants
  Abdominal Pain: Not reported | 18
  Abdominal Pain: Grade 1-mild | 2
  Abdominal Pain: Grade 2-moderate | 1
  Abdominal Pain: Grade 3-severe | 0
  Anemia: Not reported | 15
  Anemia: Grade 1-mild | 2
  Anemia: Grade 2-moderate | 4
  Anemia: Grade 3-severe | 0
  Anorexia: Not reported | 19
  Anorexia: Grade 1-mild | 2
  Anorexia: Grade 2-moderate | 0
  Anorexia: Grade 3-severe | 0
  Bladder spasm: Not reported | 20
  Bladder spasm: Grade 1-mild | 0
  Bladder spasm: Grade 2-moderate | 1
  Bladder spasm: Grade 3-severe | 0
  Bloating: Not reported | 20
  Bloating: Grade 1-mild | 1
  Bloating: Grade 2-moderate | 0
  Bloating: Grade 3-severe | 0
  Constipation: Not reported | 20
  Constipation: Grade 1-mild | 1
  Constipation: Grade 2-moderate | 0
  Constipation: Grade 3-severe | 0
  Cystitis noninfective: Not reported | 20
  Cystitis noninfective: Grade 1-mild | 1
  Cystitis noninfective: Grade 2-moderate | 0
  Cystitis noninfective: Grade 3-severe | 0
  Dermatitis radiation: Not reported | 12
  Dermatitis radiation: Grade 1-mild | 7
  Dermatitis radiation: Grade 2-moderate | 2
  Dermatitis radiation: Grade 3-severe | 0
  Diarrhea: Not reported | 6
  Diarrhea: Grade 1-mild | 10
  Diarrhea: Grade 2-moderate | 3
  Diarrhea: Grade 3-severe | 2
  Fatigue: Not reported | 3
  Fatigue: Grade 1-mild | 12
  Fatigue: Grade 2-moderate | 6
  Fatigue: Grade 3-severe | 0
  Flatulence: Not reported | 20
  Flatulence: Grade 1-mild | 1
  Flatulence: Grade 2-moderate | 0
  Flatulence: Grade 3-severe | 0
  Gastrointestinal disorders - Other, specify: Not reported | 18
  Gastrointestinal disorders - Other, specify: Grade 1-mild | 2
  Gastrointestinal disorders - Other, specify: Grade 2-moderate | 1
  Gastrointestinal disorders - Other, specify: Grade 3-severe | 0
  Hematuria: Not reported | 20
  Hematuria: Grade 1-mild | 1
  Hematuria: Grade 2-moderate | 0
  Hematuria: Grade 3-severe | 0
  Hypokalemia: Not reported | 20
  Hypokalemia: Grade 1-mild | 1
  Hypokalemia: Grade 2-moderate | 0
  Hypokalemia: Grade 3-severe | 0
  Infections and infestations - Other, specify: Not reported | 20
  Infections and infestations - Other, specify: Grade 1-mild | 0
  Infections and infestations - Other, specify: Grade 2-moderate | 1
  Infections and infestations - Other, specify: Grade 3-severe | 0
  Lymphocyte count decreased: Not reported | 12
  Lymphocyte count decreased: Grade 1-mild | 1
  Lymphocyte count decreased: Grade 2-moderate | 4
  Lymphocyte count decreased: Grade 3-severe | 4
  Nausea: Not reported | 8
  Nausea: Grade 1-mild | 11
  Nausea: Grade 2-moderate | 2
  Nausea: Grade 3-severe | 0
  Neutrophil count decreased: Not reported | 20
  Neutrophil count decreased: Grade 1-mild | 0
  Neutrophil count decreased: Grade 2-moderate | 0
  Neutrophil count decreased: Grade 3-severe | 1
  Pain: Not reported | 20
  Pain: Grade 1-mild | 1
  Pain: Grade 2-moderate | 0
  Pain: Grade 3-severe | 0
  Pelvic pain: Not reported | 20
  Pelvic pain: Grade 1-mild | 1
  Pelvic pain: Grade 2-moderate | 0
  Pelvic pain: Grade 3-severe | 0
  Platelet count decreased: Not reported | 15
  Platelet count decreased: Grade 1-mild | 3
  Platelet count decreased: Grade 2-moderate | 3
  Platelet count decreased: Grade 3-severe | 0
  Proctitis: Not reported | 18
  Proctitis: Grade 1-mild | 1
  Proctitis: Grade 2-moderate | 1
  Proctitis: Grade 3-severe | 1
  Proteinuria: Not reported | 20
  Proteinuria: Grade 1-mild | 1
  Proteinuria: Grade 2-moderate | 0
  Proteinuria: Grade 3-severe | 0
  Pruritis: Not reported | 20
  Pruritis: Grade 1-mild | 1
  Pruritis: Grade 2-moderate | 0
  Pruritis: Grade 3-severe | 0
  Rectal hemorrhage: Not reported | 19
  Rectal hemorrhage: Grade 1-mild | 2
  Rectal hemorrhage: Grade 2-moderate | 0
  Rectal hemorrhage: Grade 3-severe | 0
  Rectal pain: Not reported | 17
  Rectal pain: Grade 1-mild | 4
  Rectal pain: Grade 2-moderate | 0
  Rectal pain: Grade 3-severe | 0
  Renal and urinary disorders - other, specify: Not reported | 18
  Renal and urinary disorders - other, specify: Grade 1-mild | 3
  Renal and urinary disorders - other, specify: Grade 2-moderate | 0
  Renal and urinary disorders - other, specify: Grade 3-severe | 0
  Reproductive system and breast disorders - other, specify: Not reported | 19
  Reproductive system and breast disorders - other, specify: Grade 1-mild | 1
  Reproductive system and breast disorders - other, specify: Grade 2-moderate | 1
  Reproductive system and breast disorders - other, specify: Grade 3-severe | 0
  Skin and subcutaneous tissue disorders - other, specify: Not reported | 18
  Skin and subcutaneous tissue disorders - other, specify: Grade 1-mild | 2
  Skin and subcutaneous tissue disorders - other, specify: Grade 2-moderate | 1
  Skin and subcutaneous tissue disorders - other, specify: Grade 3-severe | 0
  Stomach pain: Not reported | 20
  Stomach pain: Grade 1-mild | 1
  Stomach pain: Grade 2-moderate | 0
  Stomach pain: Grade 3-severe | 0
  Superficial thrombophlebitis: Not reported | 20
  Superficial thrombophlebitis: Grade 1-mild | 0
  Superficial thrombophlebitis: Grade 2-moderate | 1
  Superficial thrombophlebitis: Grade 3-severe | 0
  Urinary frequency: Not reported | 17
  Urinary frequency: Grade 1-mild | 4
  Urinary frequency: Grade 2-moderate | 0
  Urinary frequency: Grade 3-severe | 0
  urinary tract infection: Not reported | 20
  urinary tract infection: Grade 1-mild | 0
  urinary tract infection: Grade 2-moderate | 1
  urinary tract infection: Grade 3-severe | 0
  Urinary tract pain: Not reported | 16
  Urinary tract pain: Grade 1-mild | 4
  Urinary tract pain: Grade 2-moderate | 1
  Urinary tract pain: Grade 3-severe | 0
  Urinary urgency: Not reported | 17
  Urinary urgency: Grade 1-mild | 4
  Urinary urgency: Grade 2-moderate | 0
  Urinary urgency: Grade 3-severe | 0
  Vaginal discharge: Not reported | 19
  Vaginal discharge: Grade 1-mild | 2
  Vaginal discharge: Grade 2-moderate | 0
  Vaginal discharge: Grade 3-severe | 0
  Vaginal dryness: Not reported | 19
  Vaginal dryness: Grade 1-mild | 2
  Vaginal dryness: Grade 2-moderate | 0
  Vaginal dryness: Grade 3-severe | 0
  Vaginal inflammation: Not reported | 19
  Vaginal inflammation: Grade 1-mild | 0
  Vaginal inflammation: Grade 2-moderate | 2
  Vaginal inflammation: Grade 3-severe | 0
  Vaginal pain: Not reported | 15
  Vaginal pain: Grade 1-mild | 6
  Vaginal pain: Grade 2-moderate | 0
  Vaginal pain: Grade 3-severe | 0
  Vomiting: Not reported | 20
  Vomiting: Grade 1-mild | 1
  Vomiting: Grade 2-moderate | 0
  Vomiting: Grade 3-severe | 0
  While blood cell decreased: Not reported | 14
  While blood cell decreased: Grade 1-mild | 5
  While blood cell decreased: Grade 2-moderate | 1
  While blood cell decreased: Grade 3-severe | 1

3. Primary Outcome: Delayed Radiation Complications
Description: Delayed complications from radiation were prospectively assessed. Below are the treatment-related late toxicities (adverse events possibly, probably, or definitely related to protocol treatment that started 6 months or later after treatment completion) that occurred on study, along with the number of participants who experienced each event at a given severity (Grade 1/mild, Grade 2/moderate, Grade 3/severe) according to the CTCAE v 4.02 (Common terminology criteria for adverse events).
Time Frame: 5 years
Population: 22 subjects enrolled, and 1 subject withdrew consent prior to treatment. The remaining 21 subjects were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Proton Radiation Therapy
Number analyzed (Participants) | 21
Participants
  Abdominal distension: Not reported | 20
  Abdominal distension: Grade 1 (mild) | 1
  Abdominal distension: Grade 2 (moderate) | 0
  Abdominal distension: Grade 3 (Severe | 0
  Abdominal pain: Not reported | 18
  Abdominal pain: Grade 1 (mild) | 2
  Abdominal pain: Grade 2 (moderate) | 1
  Abdominal pain: Grade 3 (Severe | 0
  Anal pain: Not reported | 20
  Anal pain: Grade 1 (mild) | 1
  Anal pain: Grade 2 (moderate) | 0
  Anal pain: Grade 3 (Severe | 0
  Anemia: Not reported | 20
  Anemia: Grade 1 (mild) | 1
  Anemia: Grade 2 (moderate) | 0
  Anemia: Grade 3 (Severe | 0
  Constipation: Not reported | 20
  Constipation: Grade 1 (mild) | 1
  Constipation: Grade 2 (moderate) | 0
  Constipation: Grade 3 (Severe | 0
  Cystitis noninfective: Not reported | 20
  Cystitis noninfective: Grade 1 (mild) | 1
  Cystitis noninfective: Grade 2 (moderate) | 0
  Cystitis noninfective: Grade 3 (Severe | 0
  Dermatitis radiation: Not reported | 20
  Dermatitis radiation: Grade 1 (mild) | 1
  Dermatitis radiation: Grade 2 (moderate) | 0
  Dermatitis radiation: Grade 3 (Severe | 0
  Diarrhea: Not reported | 16
  Diarrhea: Grade 1 (mild) | 4
  Diarrhea: Grade 2 (moderate) | 1
  Diarrhea: Grade 3 (Severe | 0
  Dry skin: Not reported | 20
  Dry skin: Grade 1 (mild) | 1
  Dry skin: Grade 2 (moderate) | 0
  Dry skin: Grade 3 (Severe | 0
  Duodenal ulcer: Not reported | 20
  Duodenal ulcer: Grade 1 (mild) | 0
  Duodenal ulcer: Grade 2 (moderate) | 1
  Duodenal ulcer: Grade 3 (Severe | 0
  Dyspareunia: Not reported | 19
  Dyspareunia: Grade 1 (mild) | 1
  Dyspareunia: Grade 2 (moderate) | 1
  Dyspareunia: Grade 3 (Severe | 0
  Edema limbs: Not reported | 19
  Edema limbs: Grade 1 (mild) | 2
  Edema limbs: Grade 2 (moderate) | 0
  Edema limbs: Grade 3 (Severe | 0
  Fatigue: Not reported | 17
  Fatigue: Grade 1 (mild) | 3
  Fatigue: Grade 2 (moderate) | 1
  Fatigue: Grade 3 (Severe | 0
  Fecal incontinence: Not reported | 15
  Fecal incontinence: Grade 1 (mild) | 6
  Fecal incontinence: Grade 2 (moderate) | 0
  Fecal incontinence: Grade 3 (Severe | 0
  Flatulence: Not reported | 20
  Flatulence: Grade 1 (mild) | 1
  Flatulence: Grade 2 (moderate) | 0
  Flatulence: Grade 3 (Severe | 0
  Gastritis: Not reported | 20
  Gastritis: Grade 1 (mild) | 0
  Gastritis: Grade 2 (moderate) | 1
  Gastritis: Grade 3 (Severe | 0
  Gastrointestinal disorders - other, specify: Not reported | 17
  Gastrointestinal disorders - other, specify: Grade 1 (mild) | 4
  Gastrointestinal disorders - other, specify: Grade 2 (moderate) | 0
  Gastrointestinal disorders - other, specify: Grade 3 (Severe | 0
  Hematuria: Not reported | 19
  Hematuria: Grade 1 (mild) | 2
  Hematuria: Grade 2 (moderate) | 0
  Hematuria: Grade 3 (Severe | 0
  Hemorrhoids: Not reported | 20
  Hemorrhoids: Grade 1 (mild) | 1
  Hemorrhoids: Grade 2 (moderate) | 0
  Hemorrhoids: Grade 3 (Severe | 0
  Libido decreased: Not reported | 20
  Libido decreased: Grade 1 (mild) | 0
  Libido decreased: Grade 2 (moderate) | 1
  Libido decreased: Grade 3 (Severe | 0
  Lymphedema: Not reported | 15
  Lymphedema: Grade 1 (mild) | 5
  Lymphedema: Grade 2 (moderate) | 0
  Lymphedema: Grade 3 (Severe | 1
  Lymphocyte count decreased: Not reported | 16
  Lymphocyte count decreased: Grade 1 (mild) | 4
  Lymphocyte count decreased: Grade 2 (moderate) | 1
  Lymphocyte count decreased: Grade 3 (Severe | 0
  Nausea: Not reported | 19
  Nausea: Grade 1 (mild) | 2
  Nausea: Grade 2 (moderate) | 0
  Nausea: Grade 3 (Severe | 0
  Paresthesia: Not reported | 20
  Paresthesia: Grade 1 (mild) | 0
  Paresthesia: Grade 2 (moderate) | 1
  Paresthesia: Grade 3 (Severe | 0
  Pelvic pain: Not reported | 18
  Pelvic pain: Grade 1 (mild) | 3
  Pelvic pain: Grade 2 (moderate) | 0
  Pelvic pain: Grade 3 (Severe | 0
  Proctitis: Not reported | 19
  Proctitis: Grade 1 (mild) | 2
  Proctitis: Grade 2 (moderate) | 0
  Proctitis: Grade 3 (Severe | 0
  Psychiatric disorders - other, specify: Not reported | 20
  Psychiatric disorders - other, specify: Grade 1 (mild) | 0
  Psychiatric disorders - other, specify: Grade 2 (moderate) | 1
  Psychiatric disorders - other, specify: Grade 3 (Severe | 0
  Rectal hemorrhage: Not reported | 20
  Rectal hemorrhage: Grade 1 (mild) | 1
  Rectal hemorrhage: Grade 2 (moderate) | 0
  Rectal hemorrhage: Grade 3 (Severe | 0
  Renal and urinary disorders - other, specify: Not reported | 18
  Renal and urinary disorders - other, specify: Grade 1 (mild) | 2
  Renal and urinary disorders - other, specify: Grade 2 (moderate) | 1
  Renal and urinary disorders - other, specify: Grade 3 (Severe | 0
  Reproductive system and breast disorders - other, specify: Not reported | 17
  Reproductive system and breast disorders - other, specify: Grade 1 (mild) | 4
  Reproductive system and breast disorders - other, specify: Grade 2 (moderate) | 0
  Reproductive system and breast disorders - other, specify: Grade 3 (Severe | 0
  Small intestinal obstruction: Not reported | 20
  Small intestinal obstruction: Grade 1 (mild) | 0
  Small intestinal obstruction: Grade 2 (moderate) | 0
  Small intestinal obstruction: Grade 3 (Severe | 1
  Telangiectasia: Not reported | 17
  Telangiectasia: Grade 1 (mild) | 4
  Telangiectasia: Grade 2 (moderate) | 0
  Telangiectasia: Grade 3 (Severe | 0
  Urinary frequency: Not reported | 17
  Urinary frequency: Grade 1 (mild) | 4
  Urinary frequency: Grade 2 (moderate) | 0
  Urinary frequency: Grade 3 (Severe | 0
  Urinary incontinence: Not reported | 19
  Urinary incontinence: Grade 1 (mild) | 2
  Urinary incontinence: Grade 2 (moderate) | 0
  Urinary incontinence: Grade 3 (Severe | 0
  Urinary retention: Not reported | 20
  Urinary retention: Grade 1 (mild) | 1
  Urinary retention: Grade 2 (moderate) | 0
  Urinary retention: Grade 3 (Severe | 0
  Urinary tract pain: Not reported | 20
  Urinary tract pain: Grade 1 (mild) | 1
  Urinary tract pain: Grade 2 (moderate) | 0
  Urinary tract pain: Grade 3 (Severe | 0
  Vaginal discharge: Not reported | 20
  Vaginal discharge: Grade 1 (mild) | 1
  Vaginal discharge: Grade 2 (moderate) | 0
  Vaginal discharge: Grade 3 (Severe | 0
  Vaginal dryness: Not reported | 17
  Vaginal dryness: Grade 1 (mild) | 3
  Vaginal dryness: Grade 2 (moderate) | 1
  Vaginal dryness: Grade 3 (Severe | 0
  Vaginal hemorrhage: Not reported | 18
  Vaginal hemorrhage: Grade 1 (mild) | 3
  Vaginal hemorrhage: Grade 2 (moderate) | 0
  Vaginal hemorrhage: Grade 3 (Severe | 0
  Vaginal inflammation: Not reported | 20
  Vaginal inflammation: Grade 1 (mild) | 1
  Vaginal inflammation: Grade 2 (moderate) | 0
  Vaginal inflammation: Grade 3 (Severe | 0
  Vaginal obstruction: Not reported | 20
  Vaginal obstruction: Grade 1 (mild) | 1
  Vaginal obstruction: Grade 2 (moderate) | 0
  Vaginal obstruction: Grade 3 (Severe | 0
  Vaginal pain: Not reported | 18
  Vaginal pain: Grade 1 (mild) | 2
  Vaginal pain: Grade 2 (moderate) | 1
  Vaginal pain: Grade 3 (Severe | 0
  Vaginal stricture: Not reported | 19
  Vaginal stricture: Grade 1 (mild) | 1
  Vaginal stricture: Grade 2 (moderate) | 1
  Vaginal stricture: Grade 3 (Severe | 0
  Vomiting: Not reported | 20
  Vomiting: Grade 1 (mild) | 1
  Vomiting: Grade 2 (moderate) | 0
  Vomiting: Grade 3 (Severe | 0
  Vulval infection: Not reported | 20
  Vulval infection: Grade 1 (mild) | 1
  Vulval infection: Grade 2 (moderate) | 0
  Vulval infection: Grade 3 (Severe | 0
  Weight gain: Not reported | 20
  Weight gain: Grade 1 (mild) | 1
  Weight gain: Grade 2 (moderate) | 0
  Weight gain: Grade 3 (Severe | 0
  White blood cell decreased: Not reported | 20
  White blood cell decreased: Grade 1 (mild) | 1
  White blood cell decreased: Grade 2 (moderate) | 0
  White blood cell decreased: Grade 3 (Severe | 0

4. Secondary Outcome: Quality of Life (QOL)
Description: The total FACT-EN/Cx scale (Functional Assessment of Cancer Therapy - Endometrial/Cervical) score was assessed at baseline and timepoints of 6 months, 1 year, 2 years, 3 years, 4 years, and 5 years to evaluate quality of life (QOL) before and after adjuvant scanning proton beam therapy.
  Unit = Scores on a scale. Subset scores are summed together to get a total score.
  Functional Assessment of Cancer Therapy - Endometrial - score range 0 - 172, with higher scores indicating a better outcome Functional Assessment of Cancer Therapy - Cervical - score range 0 - 168, with higher scores indicating a better outcome
Time Frame: Baseline, 6 months, 1 year, 2 years, 3 years, 4 years, and 5 years
Population: 22 patients were enrolled, 1 of whom withdrew consent prior to study treatment. The remaining 21 subjects were analyzed.
Measure: Mean (Standard Deviation); unit: total score on FACT-EN/Cx scale
Arm/Group | Proton Radiation Therapy
Number analyzed (Participants) | 21
total score on FACT-EN/Cx scale
  Baseline | 128.67 (25.88)
  6 months | 133.47 (29.55)
  1 year | 131.53 (27.49)
  2 years | 133.65 (25.71)
  3 years | 139.13 (24.62)
  4 years | 142.88 (21.93)
  5 years | 149.39 (14.30)

5. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS is defined as the duration of time from start of treatment to time of objective disease progression at any site as detected by symptomatic recurrence or routine surveillance follow-up physical examination/imaging, or death from any cause.
Time Frame: 12 months, 24 months, 36 months, 48 months, and 60 months
Population: 22 patients were enrolled, 1 of whom withdrew prior to study treatment. The remaining 21 patients were included in this analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Proton Radiation Therapy
Number analyzed (Participants) | 21
percentage of participants
  12 months post treatment completion | 85.7 [62.0 to 95.2]
  24 months post treatment completion | 80.7 [56.3 to 92.3]
  36 months post treatment completion | 75.6 [50.9 to 89.1]
  48 months post treatment completion | 75.6 [50.9 to 89.1]
  60 months post treatment completion | 75.6 [50.9 to 89.1]

ADVERSE EVENTS:
Time Frame: Adverse events will be collected and reported from initiation of study treatment until 60 months after the last dose of study medication/radiation treatment (5 years). This was assessed every 3 months years 1-2 post-treatment, every 4 months year 3, and every 6 months until 5 years from the end of the last dose of radiation.
Arm/Group | Proton Radiation Therapy
All-Cause Mortality (participants affected / at risk) | 0/21
Serious Adverse Events (participants affected / at risk) | 0/21
Other Adverse Events (participants affected / at risk) | 21/21
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Proton Radiation Therapy (N=21)
Abdominal distension (Gastrointestinal disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 12
Acute kidney injury (Renal and urinary disorders) | 2
Agitation (Psychiatric disorders) | 2
Alkaline phosphatase increased (Investigations) | 6
Allergic reaction (Immune system disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 5
Amnesia (Nervous system disorders) | 1
Anal hemorrhage (Gastrointestinal disorders) | 1
Anal pain (Gastrointestinal disorders) | 1
Anemia (Blood and lymphatic system disorders) | 13
Anorexia (Metabolism and nutrition disorders) | 7
Anxiety (Psychiatric disorders) | 9
Apnea (Respiratory, thoracic and mediastinal disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 5
Ascites (Gastrointestinal disorders) | 2
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1
Atrial fibrillation (Cardiac disorders) | 2
Atrial flutter (Cardiac disorders) | 1
Autoimmune disorder (Immune system disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 9
Bladder spasm (Renal and urinary disorders) | 1
Bloating (Gastrointestinal disorders) | 5
Blood and lymphatic system disorders - Other, specify: Iron deficiency (Blood and lymphatic system disorders) | 1
Blood and lymphatic system disorders - Other, specify: Mucosal hyperemia (Blood and lymphatic system disorders) | 1
Blood corticotrophin decreased (Investigations) | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 3
Breast pain (Reproductive system and breast disorders) | 2
Bruising (Injury, poisoning and procedural complications) | 5
Buttock pain (Musculoskeletal and connective tissue disorders) | 1
Cardiac disorders - Other, specify: Carotid bruit (Cardiac disorders) | 1
Cardiac disorders - Other, specify: Abdominal aortic pulsation (Cardiac disorders) | 1
Cardiac disorders - Other, specify: Dilated cardiomyopathy (Cardiac disorders) | 1
Cardiac disorders - Other, specify: systolic murmur (Cardiac disorders) | 2
Cardiac disorders - Other, specify (Cardiac disorders) | 1
Cataract (Eye disorders) | 2
Chest pain - cardiac (Cardiac disorders) | 1
Chills (General disorders) | 3
Cholecystitis (Hepatobiliary disorders) | 1
Cholesterol high (Investigations) | 2
Colitis (Gastrointestinal disorders) | 1
Confusion (Psychiatric disorders) | 3
Constipation (Gastrointestinal disorders) | 19
Cough (Respiratory, thoracic and mediastinal disorders) | 7
Cystitis noninfective (Renal and urinary disorders) | 2
Dehydration (Metabolism and nutrition disorders) | 3
Dental caries (Gastrointestinal disorders) | 1
Depression (Psychiatric disorders) | 5
Dermatitis radiation (Injury, poisoning and procedural complications) | 10
Diarrhea (Gastrointestinal disorders) | 16
Dizziness (Nervous system disorders) | 6
Dry mouth (Gastrointestinal disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 4
Duodenal hemorrhage (Gastrointestinal disorders) | 2
Duodenal ulcer (Gastrointestinal disorders) | 1
Dysgeusia (Nervous system disorders) | 2
Dyspareunia (Reproductive system and breast disorders) | 3
Dyspepsia (Gastrointestinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 10
Ear pain (Ear and labyrinth disorders) | 2
Edema face (General disorders) | 1
Edema limbs (General disorders) | 12
Endocrine disorders - Other, specify: bilateral small hypoechoic nodules; benign appearance (Endocrine disorders) | 1
Endocrine disorders - Other, specify: Multinodular goiter (Endocrine disorders) | 1
Enterocolitis (Gastrointestinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Erythema multiforme (Skin and subcutaneous tissue disorders) | 4
Eye disorders - Other, specify: exopthalmos (Eye disorders) | 1
Eye disorders - Other, specify: Left upper lid pain - swollen, crusty discharge (Eye disorders) | 1
Eye disorders - Other, specify: hordeolum externum of left upper eyelid (Eye disorders) | 1
Eye disorders - Other, specify: pain and swelling in Right upper eyelid (Eye disorders) | 1
Eye disorders - Other, specify: pathologic myopia (Eye disorders) | 1
Eye disorders - Other, specify: asthenopia (Eye disorders) | 1
Eye disorders - Other, specify: meibomian gland dysfunction (Eye disorders) | 1
Eye pain (Eye disorders) | 2
Fall (Injury, poisoning and procedural complications) | 3
Fatigue (General disorders) | 20
Fecal incontinence (Gastrointestinal disorders) | 11
Fever (General disorders) | 4
Flatulence (Gastrointestinal disorders) | 7
Floaters (Eye disorders) | 1
Flu like symptoms (General disorders) | 1
Flushing (Vascular disorders) | 1
Fracture (Injury, poisoning and procedural complications) | 1
Gait disturbance (General disorders) | 3
Gastritis (Gastrointestinal disorders) | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 7
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 3
Gastrointestinal disorders - Other, specify: history of crohn's disease (Gastrointestinal disorders) | 1
Gastrointestinal disorders - Other, specify: small bowel obstruction (Gastrointestinal disorders) | 1
Gastrointestinal disorders - Other, specify: abdominal spasms (Gastrointestinal disorders) | 1
Gastrointestinal disorders - Other, specify: Rectal urgency (Gastrointestinal disorders) | 1
Gastrointestinal disorders - Other, specify: Diverticulosis (Gastrointestinal disorders) | 2
Gastrointestinal disorders - Other, specify: Rectal discharge (Gastrointestinal disorders) | 1
Gastrointestinal disorders - Other, specify: Abdominal discomfort secondary to oral contrast agent (Gastrointestinal disorders) | 1
Gastrointestinal disorders - Other, specify: Hiatal hernia (Gastrointestinal disorders) | 1
Gastrointestinal disorders - Other, specify: Melena (Gastrointestinal disorders) | 1
Gastrointestinal disorders - Other, specify: Hematochezia (Gastrointestinal disorders) | 1
Gastrointestinal disorders - Other, specify: Rectocele (Gastrointestinal disorders) | 1
Gastrointestinal disorders - Other, specify: Irritable bowel syndrome (Gastrointestinal disorders) | 1
Gastrointestinal disorders - Other, specify: Rectal urgency (Gastrointestinal disorders) | 2
Gastrointestinal disorders - Other, specify: Bowel urgency (Gastrointestinal disorders) | 1
Gastrointestinal disorders - Other, specify: increased frequency of bowel movements (Gastrointestinal disorders) | 1
General disorders and administration site conditions - Other, specify: Diaphoresis (General disorders) | 1
General disorders and administration site conditions - Other, specify: lesion on finger (General disorders) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 3
Glaucoma (Eye disorders) | 2
Gum infection (Infections and infestations) | 1
Hallucinations (Psychiatric disorders) | 1
Headache (Nervous system disorders) | 7
Hearing impaired (Ear and labyrinth disorders) | 3
Heart failure (Cardiac disorders) | 1
Hematuria (Renal and urinary disorders) | 3
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 2
Hemorrhoids (Gastrointestinal disorders) | 7
Hepatobiliary disorders - Other, specify: cholelithisasis (Hepatobiliary disorders) | 1
Hirsutism (Skin and subcutaneous tissue disorders) | 2
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 2
Hot flashes (Vascular disorders) | 3
Hyperglycemia (Metabolism and nutrition disorders) | 7
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3
Hyperkalemia (Metabolism and nutrition disorders) | 2
Hypertension (Vascular disorders) | 4
Hyperthyroidism (Endocrine disorders) | 2
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 1
Hypocalcemia (Metabolism and nutrition disorders) | 4
Hypokalemia (Metabolism and nutrition disorders) | 2
Hypomagnesemia (Metabolism and nutrition disorders) | 3
Hyponatremia (Metabolism and nutrition disorders) | 2
Hypophosphatemia (Metabolism and nutrition disorders) | 1
Hypotension (Vascular disorders) | 2
Hypothyroidism (Endocrine disorders) | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3
Infections and infestations - Other, specify: herpes simplex virus (Infections and infestations) | 1
Infections and infestations - Other, specify: tooth infection (Infections and infestations) | 1
Infections and infestations - Other, specify: yeast infection (Infections and infestations) | 1
Injury, poisoning and procedural complications - Other, specify: rotator cuff tear (Injury, poisoning and procedural complications) | 1
Injury, poisoning and procedural complications - Other, specify: port site pain (Injury, poisoning and procedural complications) | 1
INR increased (Investigations) | 1
Insomnia (Psychiatric disorders) | 6
Irritability (General disorders) | 1
Kidney infection (Infections and infestations) | 1
Libido decreased (Psychiatric disorders) | 3
Lip infection (Infections and infestations) | 1
Localized edema (General disorders) | 1
Lymphedema (Vascular disorders) | 7
Lymphocyte count decreased (Investigations) | 13
Metabolism and nutrition disorders - Other, specify: Insulin resistance (Metabolism and nutrition disorders) | 1
Metabolism and nutrition disorders - Other, specify: lactic acidosis (Metabolism and nutrition disorders) | 1
Metabolism and nutrition disorders - Other, specify: vitamin D deficiency (Metabolism and nutrition disorders) | 1
Musculoskeletal and connective tissue disorder - Other, specify: hip pain (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal and connective tissue disorder - Other, specify: knee pain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal and connective tissue disorder - Other, specify: plantar lesion (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal and connective tissue disorder - Other, specify: Soft bulging when standing up (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal and connective tissue disorder - Other, specify: degenerative disc disease (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal and connective tissue disorder - Other, specify: finger pain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal and connective tissue disorder - Other, specify: subacromial spur w/ tendinopathy (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal and connective tissue disorder - Other, specify: hyperreflexia (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal and connective tissue disorder - Other, specify: Sciatica (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal and connective tissue disorder - Other, specify: Fibromyalgia (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal and connective tissue disorder - Other, specify: osteitis deformans (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal and connective tissue disorder - Other, specify: Musculoskeletal deformity (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 6
Nail discoloration (Skin and subcutaneous tissue disorders) | 1
Nail infection (Infections and infestations) | 1
Nail loss (Skin and subcutaneous tissue disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4
Nausea (Gastrointestinal disorders) | 18
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify: Vascular polyp (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify: Baker's cyst (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify: Cyst (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify: Ganglion cyst (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Nervous system disorders - Other, specify: hyperreflexia (Nervous system disorders) | 1
Nervous system disorders - Other, specify (Nervous system disorders) | 1
Nervous system disorders - Other, specify: Carpal tunnel syndrome (Nervous system disorders) | 1
Neuralgia (Nervous system disorders) | 1
Neutrophil count decreased (Investigations) | 2
Non-cardiac chest pain (General disorders) | 3
Obesity (Metabolism and nutrition disorders) | 3
Oral pain (Gastrointestinal disorders) | 1
Pain (General disorders) | 10
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6
Palpitations (Cardiac disorders) | 4
Paresthesia (Nervous system disorders) | 3
Pelvic pain (Reproductive system and breast disorders) | 7
Periorbital edema (Skin and subcutaneous tissue disorders) | 1
Peripheral motor neuropathy (Nervous system disorders) | 2
Peripheral sensory neuropathy (Nervous system disorders) | 12
Pharyngitis (Infections and infestations) | 1
Photosensitivity (Skin and subcutaneous tissue disorders) | 1
Platelet count decreased (Investigations) | 7
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 4
Premature menopause (Reproductive system and breast disorders) | 2
Proctitis (Gastrointestinal disorders) | 5
Productive cough (Respiratory, thoracic and mediastinal disorders) | 4
Proteinuria (Renal and urinary disorders) | 4
Pruritus (Skin and subcutaneous tissue disorders) | 3
Psychiatric disorders - Other, specify: PTSD (Psychiatric disorders) | 1
Psychiatric disorders - Other, specify: Recent cognitive struggles, sleep disruption and sadness. (Psychiatric disorders) | 1
Psychiatric disorders - Other, specify: ADHD (Psychiatric disorders) | 1
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3
Rectal hemorrhage (Gastrointestinal disorders) | 5
Rectal mucositis (Gastrointestinal disorders) | 1
Rectal pain (Gastrointestinal disorders) | 6
Renal and urinary disorders - Other, specify: Dysuria (Renal and urinary disorders) | 4
Renal and urinary disorders - Other, specify: Bladder pressure and urinary frequency (Renal and urinary disorders) | 1
Renal and urinary disorders - Other, specify: Mons swelling (Renal and urinary disorders) | 1
Renal and urinary disorders - Other, specify: cytocele (Renal and urinary disorders) | 1
Renal and urinary disorders - Other, specify: Urinary leakage (Renal and urinary disorders) | 1
Renal and urinary disorders - Other, specify: Suprapubic pressure and discomfort with urination (Renal and urinary disorders) | 1
Reproductive system and breast disorders - Other, specify: changes to vaginal mucosa (Reproductive system and breast disorders) | 1
Reproductive system and breast disorders - Other, specify: Synechiae in vagina (Reproductive system and breast disorders) | 1
Reproductive system and breast disorders - Other, specify: radiation changes in vagina (Reproductive system and breast disorders) | 2
Reproductive system and breast disorders - Other, specify: Vaginal bleeding (Reproductive system and breast disorders) | 1
Reproductive system and breast disorders - Other, specify: Radiation stigmata (Reproductive system and breast disorders) | 2
Reproductive system and breast disorders - Other, specify: Yeast infection (Reproductive system and breast disorders) | 1
Reproductive system and breast disorders - Other, specify: Vaginal discharge discoloration (Reproductive system and breast disorders) | 1
Reproductive system and breast disorders - Other, specify: Vaginitis (Reproductive system and breast disorders) | 1
Reproductive system and breast disorders - Other, specify: Vaginal bleeding during intercourse (Reproductive system and breast disorders) | 1
Reproductive system and breast disorders - Other, specify: Post-coital bleeding (Reproductive system and breast disorders) | 1
Reproductive system and breast disorders - Other, specify: Perineal erythema (Reproductive system and breast disorders) | 1
Reproductive system and breast disorders - Other, specify: Vaginal atrophy (Reproductive system and breast disorders) | 2
Reproductive system and breast disorders - Other, specify: Vaginal mucosa atrophy (Reproductive system and breast disorders) | 1
Reproductive system and breast disorders - Other, specify: Mons pubis swelling, pressure, discomfort (Reproductive system and breast disorders) | 1
Reproductive system and breast disorders - Other, specify: Mild hyperemia of vagina (Reproductive system and breast disorders) | 1
Reproductive system and breast disorders - Other, specify: Radiation changes/erythema at the cuff (Reproductive system and breast disorders) | 1
Reproductive system and breast disorders - Other, specify (Reproductive system and breast disorders) | 1
Reproductive system and breast disorders - Other, specify: Vaginal burning (Reproductive system and breast disorders) | 2
Reproductive system and breast disorders - Other, specify: Radiation fibrosis of vaginal rugae (Reproductive system and breast disorders) | 1
Reproductive system and breast disorders - Other, specify: Enlarged veins R labial vulvar region (Reproductive system and breast disorders) | 1
Reproductive system and breast disorders - Other, specify: Sphincter tone decreased (Reproductive system and breast disorders) | 1
Reproductive system and breast disorders - Other, specify: vulva lesions (Reproductive system and breast disorders) | 1
Respiratory, thoracic and mediastinal disorders - Other, specify: Tachypnea (Respiratory, thoracic and mediastinal disorders) | 1
Retinal tear (Eye disorders) | 1
Sepsis (Infections and infestations) | 1
Sinus bradycardia (Cardiac disorders) | 1
Sinus pain (Nervous system disorders) | 1
Sinus tachycardia (Cardiac disorders) | 1
Skin and subcutaneous tissue disorders - Other, specify: Ingrown toenail (Skin and subcutaneous tissue disorders) | 1
Skin and subcutaneous tissue disorders - Other, specify: rash (Skin and subcutaneous tissue disorders) | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1
Skin induration (Skin and subcutaneous tissue disorders) | 2
Skin infection (Infections and infestations) | 4
Skin/subcutaneous tissue disorders; Other, specify: Rash on inner surface of elbows (Skin and subcutaneous tissue disorders) | 1
Skin/subcutaneous tissue disorders; Other: Erythematous macular rash, venous stasis dermatitis (Skin and subcutaneous tissue disorders) | 1
Skin/subcutaneous tissue disorders; Other, specify: Seborrheic keratosis (Skin and subcutaneous tissue disorders) | 1
Skin/subcutaneous tissue disorders; Other, specify: Slight pinkness on chest (Skin and subcutaneous tissue disorders) | 1
Skin/subcutaneous tissue disorders; Other, specify: Skin tag swollen and painful left axilla (Skin and subcutaneous tissue disorders) | 1
Skin/subcutaneous tissue disorders; Other, specify: Yeast dermatitis (Skin and subcutaneous tissue disorders) | 1
Skin/subcutaneous tissue disorders; Other, specify: perineal itching (Skin and subcutaneous tissue disorders) | 1
Skin/subcutaneous tissue disorders; Other, specify: itchy rash on arms (Skin and subcutaneous tissue disorders) | 1
Skin/subcutaneous tissue disorders; Other, specify: Perineal irritation (Skin and subcutaneous tissue disorders) | 1
Skin/subcutaneous tissue disorders; Other, specify: Onychocryptosis (Skin and subcutaneous tissue disorders) | 1
Skin/subcutaneous tissue disorders; Other, specify: Erythema (Skin and subcutaneous tissue disorders) | 2
Skin/subcutaneous tissue disorders; Other, specify: lichen planus (Skin and subcutaneous tissue disorders) | 1
Skin/subcutaneous tissue disorders; Other, specify: Eczema (Skin and subcutaneous tissue disorders) | 1
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 4
Small intestinal obstruction (Gastrointestinal disorders) | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 4
Spasticity (Nervous system disorders) | 1
Spinal fracture (Injury, poisoning and procedural complications) | 1
Stomach pain (Gastrointestinal disorders) | 2
Suicidal ideation (Psychiatric disorders) | 1
Superficial thrombophlebitis (Vascular disorders) | 2
Surgical and medical procedures - Other, specify: Laparoscopic gastric bypass surgery (Surgical and medical procedures) | 1
Syncope (Nervous system disorders) | 1
Telangiectasia (Skin and subcutaneous tissue disorders) | 6
Thromboembolic event (Vascular disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 1
Tooth infection (Infections and infestations) | 1
Tremor (Nervous system disorders) | 2
Upper respiratory infection (Infections and infestations) | 3
Urinary frequency (Renal and urinary disorders) | 13
Urinary incontinence (Renal and urinary disorders) | 9
Urinary retention (Renal and urinary disorders) | 1
Urinary tract infection (Infections and infestations) | 6
Urinary tract pain (Renal and urinary disorders) | 9
Urinary urgency (Renal and urinary disorders) | 7
Vaginal discharge (Reproductive system and breast disorders) | 5
Vaginal dryness (Reproductive system and breast disorders) | 6
Vaginal hemorrhage (Reproductive system and breast disorders) | 8
Vaginal infection (Infections and infestations) | 1
Vaginal inflammation (Reproductive system and breast disorders) | 3
Vaginal obstruction (Reproductive system and breast disorders) | 1
Vaginal pain (Reproductive system and breast disorders) | 12
Vaginal stricture (Reproductive system and breast disorders) | 3
Vascular access complication (Injury, poisoning and procedural complications) | 1
Vascular disorders - Other, specify: Peripheral artery disease (Vascular disorders) | 1
Vascular disorders - Other, specify: Varicose veins (Vascular disorders) | 2
Vascular disorders - Other, specify: Venous incompetence (Vascular disorders) | 1
Vertigo (Ear and labyrinth disorders) | 2
Vomiting (Gastrointestinal disorders) | 9
Vulval infection (Infections and infestations) | 3
Weight gain (Investigations) | 5
Weight loss (Investigations) | 7
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2
White blood cell decreased (Investigations) | 8
Wound infection (Infections and infestations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-10-09): https://cdn.clinicaltrials.gov/large-docs/40/NCT01600040/Prot_SAP_000.pdf
  • Informed Consent Form (2019-10-28): https://cdn.clinicaltrials.gov/large-docs/40/NCT01600040/ICF_001.pdf